CLINICAL TRIAL: NCT05366478
Title: A Single-Arm, Open-Label, Exploratory Study to Evaluate Safety and Efficacy of LM103 Injection in the Treatment of Advanced Solid Tumors
Brief Title: A Clinical Study of LM103 Injection in the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou BlueHorse Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIL-2021001
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Melanoma; Non Small Cell Lung Cancer; Cervical Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous tumor infiltrating lymphocytes (TILs) (Experimental): In vitro expanded autologous TILs will be infused i.v. to patients with advanced solid tumors
  Interventions: Drug: Autologous tumor infiltrating lymphocytes (TILs)

INTERVENTIONS:
Drug: Autologous tumor infiltrating lymphocytes (TILs) — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepletion, patients will be infused with LM103 Injection followed by IL-2.
  Other Names: LM103

SUMMARY:
This is a single-arm, open-label, exploratory study to evaluate safety and efficacy of LM103 Injection in patients with advanced solid tumors. The purpose of this study is to evaluate the safety and tolerability, antitumor activity and immunoreactivity.

DETAILED DESCRIPTION:
This is an investigator initiated , single-arm, open-label ,exploratory study of LM103 Injection in patients with advanced solid tumors. Expanded TILs will be transferred to the patient after chemotherapy with cyclophosphamide and fludarabine. LM103 will be administered as a single dose on day 1. TIL transfer will be combined with IL-2 treatment. This study is planned to enroll 9-15 patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. AJCC (V8) stage III or IV melanoma, non-small cell lung cancer, cervical cancer and other solid tumors (confirmed by histology) for which existing treatment is ineffective or without standard treatment;
2. The patient has residual lesions that can be used for surgical resection (>1.5cm3) or biopsy (>1.5cm3) and measurable after resection for TIL collection and efficacy evaluation;
3. Laboratory inspection index requirements:

   * Blood routine: lymphocyte ratio > 20%; neutrophil count > 1.0 × 10^9/L; white blood cells > 3.0 × 10^9/L; platelets > 100 × 10^9/L; hemoglobin > 80 g/ L;
   * Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ upper limit of normal x 2.5, if there is liver metastasis ≤ upper limit of normal x 5; alkaline phosphatase (ALP) ≤ upper limit of normal x 2.5; total gallbladder Red pigment (TBIL)≤normal upper limit×1.5;
   * Renal function: urea ≤ upper limit of normal × 1.5; creatinine (Cr) ≤ upper limit of normal × 1.5;
4. Left ventricular ejection fraction (LVEF) ≥ 50%;
5. ECOG physical condition is 0 or 1;
6. The expected survival time is more than 3 months;

Exclusion Criteria:

1. Suffering from active or previous autoimmune diseases ;
2. Severe liver and kidney dysfunction, severe heart disease, coagulation dysfunction, and hematopoietic dysfunction;
3. Combined with severe infection or persistent infection and cannot be effectively controlled;
4. Central nervous system metastasis and/or cancerous meningitis;
5. With uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage;
6. Requires systemic steroid therapy;
7. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HbcAb); positive for hepatitis C virus (HCV) antibody; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Up to 1 years
  Adverse events are graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
Number of Participants With Objective Response | Up to 2 years
  Participants displaying objective response associated with the treatment regimen per Response Evaluation Criteria in Solid Tumors (RECIST v.1.1). The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
Disease Control Rate (DCR） | Up to 2 years
  Percentage of patients that meet CR, PR and SD criteria set in this study according to RECIST v1.1：
Progression-Free Survival (PFS) | Up to 2 years
  The time length between TIL infusion and confirmed subsequent disease progression according to RECIST 1.1
The changes of the immunoreactivity during treatment | Up to 2 years
  The changes from baseline of systemic immune Response markers: peripheral blood lymphocyte subtypes counts, cytokine, antigen-specific T-lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Fenge Le, Ph.D, Principal Investigator — Tianjin Beichen Hospital
Locations (1):
- Tianjin Beichen Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li F, Wang Y, Yan J, Wu H, Du X, Feng W, Zhang X, Xue Y, Wang H, Liu W. Autologous Tumor-Infiltrating Lymphocyte Mono-Therapy Can Rapidly Shrank Tumor in Asian Patient with Stage III/IV Cervical Cancer: Two Cases Report. Int J Womens Health. 2024 Jan 9;16:31-39. doi: 10.2147/IJWH.S446768. eCollection 2024. PMID 38222312